CLINICAL TRIAL: NCT01816165
Title: Role of Lipotoxicity in Insulin Resistance, Vascular, and Mitochondrial Dysfunction in Type 1 Diabetes
Brief Title: Effects of Acipimox on Insulin Action, Vascular Function, and Muscle Function in Type 1 Diabetes
Acronym: AcT1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11-0649; 6181 (Other: CTRC)
Record Dates: First submitted 2012-06-13; First posted 2013-03-22 (Estimated); Results first posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; insulin; blood vessel; type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — acipimox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acipimox (Experimental): Drug: acipimox
  Interventions: Drug: Acipimox
- Placebo (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acipimox — Subjects will take acipimox 250mg by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day.
  Other Names: Olbetam
  Arms: Acipimox
Drug: Placebo — Subjects will take placebo by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day
  Arms: Placebo

SUMMARY:
Insulin resistance (IR) is an important contributor to increased cardiovascular disease risk in type 1 diabetes (T1D). Non-esterified fatty acid elevation is a significant contributor to IR in T1D and may be a target of intervention. The hypothesis of the study is that isolated fatty acid lowering with acipimox will improve insulin action and blood vessel function and have the benefit of reducing mitochondrial oxidant generation and improving mitochondrial function in T1D. Targeting IR through fatty acid lowering is a novel approach to T1D treatment that may significantly improve current management of TID and of cardiovascular disease (CVD) risk in this high risk population.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, with and without type 1 diabetes between 25-59 years of age,
2. HbA1c 6.0-9.5 (T1D only),
3. Subjects who are willing to commit to:

   * 14 days of prescribed diet,
   * two 44 hour inpatient stays, and
   * two muscle biopsies.

Exclusion Criteria:

1. Any comorbid condition associated with inflammation, insulin resistance, or dyslipidemia,
2. Tobacco use,
3. Pregnancy,
4. Steroid use,
5. Scheduled physical activity >3 days a week,
6. Angina or any other cardiovascular or pulmonary disease,
7. History of chronic obstructive pulmonary disease or asthma,
8. Systolic blood pressure >190 at rest or >250 with exercise, or
9. Diastolic pressure >95 at rest, or >105 with exercise,
10. Proteinuria (urine protein >200 mg/dl), or
11. Creatinine > 2 mg/dl, suggestive of severe renal disease,
12. Severe Proliferative retinopathy,
13. Niacin treatment,
14. History of peptic ulcers,
15. History of hereditary angioedema, and
16. C1 esterase deficiency.

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06-24 (Actual); Study Completion 2015-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Schauer, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants (7 withdrawals, 3 screen fails) were excluded from the study after enrollment, but prior to beginning the study. One T1D acipimox to placebo was withdrawn during the acipimox phase due to an SAE.
Groups:
- Participants With T1 Diabetes: Acipimox, Then Placebo; Participants Without T1 Diabetes: Acipimox, Then Placebo: Subjects will take acipimox 250mg by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day, followed by placebo by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day.
- Participants With T1 Diabetes: Placebo, Then Acipimox; Participants Without T1 Diabetes: Placebo, Then Acipimox: Subjects will take placebo by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day, followed by acipimox 250mg by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day.
Period: Overall Study
Arm/Group | Participants With T1 Diabetes: Acipimox, Then Placebo | Participants Without T1 Diabetes: Acipimox, Then Placebo | Participants With T1 Diabetes: Placebo, Then Acipimox | Participants Without T1 Diabetes: Placebo, Then Acipimox
Started | 5 | 4 | 5 | 4
Completed Intervention 1 | 4 | 4 | 5 | 4
Completed ~2 Week Washout | 4 | 4 | 5 | 4
Started Second Intervention | 4 | 4 | 5 | 4
Completed | 4 | 4 | 5 | 4
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants With T1 Diabetes: Acipimox, Then Placebo: Subjects will take acipimox 250mg by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day, followed by placebo by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day.
  Placebo, then Acipimox :Subjects will take placebo by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day, followed by acipimox 250mg by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day.
- All Participants Without T1 Diabetes: Placebo, then Acipimox :Subjects will take placebo by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day, followed by acipimox 250mg by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day.
  Acipimox, Then Placebo: Subjects will take acipimox 250mg by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day, followed by placebo by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day.
- Total: Total of all reporting groups
Arm/Group | All Participants With T1 Diabetes | All Participants Without T1 Diabetes | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 10 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity: M-value From Hyperinsulinemic Euglycemia Clamp Study
Description: Evaluate the impact of Non esterified fatty acid (NEFA)-lowering on insulin sensitivity in T1D versus non-DM. Glucose infusion rate is reported normalized to lean body weight in kg and to final insulin concentration.
  The unit of measure reflects the rate at which glucose needs to be infused to maintain a normal blood sugar in the setting of a given serum insulin level from an insulin infusion. As such, a higher number means more glucose was needed and indicates greater sensitivity to insulin.
Time Frame: day 8 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: 1 participant in the T1 Diabetes groups was excluded from the analysis because data was only collected in the Acipimox phase and matching Placebo data would have been required for comparison.
Measure: Mean (Standard Deviation); unit: mg/kg*minute*microIU/mL*100
Groups:
- T1 Diabetes, Acipimox; No T1 Diabetes, Acipimox: Drug: acipimox
  Acipimox: Subjects will take acipimox 250mg by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day.
- T1 Diabetes, Placebo; No T1 Diabetes, Placebo: Drug: Placebo
  Placebo: Subjects will take placebo by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 8
mg/kg*minute*microIU/mL*100 | 4.65 (1.52) | 3.67 (1.45) | 8.8 (3.04) | 9.05 (2.88)

2. Primary Outcome: 24 Hour Mean Fatty Acid Levels
Description: Assesses whether fatty acid level is consistently lowered by acipimox. Mean of fatty acid levels measured 22 times over 24 hours (hourly except 0100 and 0300 hours).
Time Frame: day 6 to 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Measure: Mean (Standard Deviation); unit: microEq/L
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 8
microEq/L | 343 (122) | 297 (56) | 298 (90) | 335 (65)

3. Primary Outcome: Percent Flow-mediated Brachial Artery Dilation
Description: To determine the effects of NEFA lowering and insulin sensitization on endothelial function. Measures percent change in brachial artery diameter with hyperemia after occlusion.
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change in BA diameter
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 8
Percent change in BA diameter | 8.21 (3.02) | 8.82 (4.40) | 5.88 (4.17) | 7.32 (4.25)

4. Primary Outcome: State 3 Mitochondrial Oxygen Consumption
Description: Measures skeletal muscle mitochondrial function and effects of acipimox thereon, carbohydrate & lipid substrates. State 3 is fully active coupled oxygen flux using PMG or PMGS (pyruvate, malate, glutamate, +/- succinate) or OCMS (octanyl carnitine, malate, +/- succinate) as substrates. FCCP is added as an uncoupler to measure maximum possible O2 flux. Higher values reflect better mitochondrial function.
Time Frame: muscle biopsy on day 7 of each weeklong intervention period; max 16 weeks post enrollment
Population: 1 participant in the T1 Diabetes groups was excluded from the analysis because data was only collected in the Acipimox phase and matching Placebo data would have been required for comparison. Another participant did not have a muscle biopsy collected (T1D, Acipimox).
Measure: Mean (Standard Deviation); unit: pmoles/mg/s
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 8 | 9 | 8 | 8
pmoles/mg/s
  PMG State 3 Oxygen Flux | 26.1 (8.3) | 24.9 (7.6) | 30.2 (9.8) | 29.7 (10.0)
  PMGS State 3 Oxygen Flux | 38.0 (11.8) | 36.9 (12.7) | 42.5 (15.0) | 42.5 (11.8)
  PMGS Uncoupled Max Oxygen Flux | 65.2 (18.4) | 62.1 (16.3) | 77.8 (26.3) | 80.2 (28.9)
  OCM State 3 Oxygen Flux | 14.0 (5.8) | 15.0 (5.6) | 18.8 (8.6) | 17.3 (4.4)
  OCMS State 3 Oxygen Flux | 38.6 (14.6) | 38.5 (11.2) | 43.8 (13.3) | 41.7 (9.9)
  OCMS Uncoupled Max Oxygen Flux | 51.8 (22.9) | 56.4 (20.0) | 80.1 (24.8) | 73.1 (18.8)

5. Secondary Outcome: Oxidative Stress and Inflammatory Markers: Interleukin 6 (IL6)
Description: Interleukin 6 (IL6)
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 8
picograms/mL | 2.8 (1.6) | 4.2 (3.2) | 2.6 (2.4) | 3.5 (1.3)

6. Secondary Outcome: Oxidative Stress and Inflammatory Markers: TNFalpha
Description: TNFalpha
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: 1 participant in the T1 Diabetes groups was excluded from the analysis because data was only collected in the Acipimox phase and matching Placebo data would have been required for comparison. Two other participants (T1D, Acipimox; No T1D Acipimox) did not have data collected.
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 8 | 9 | 7 | 8
picograms/mL | 1.76 (1.08) | 1.71 (.80) | 1.56 (.95) | .91 (.46)

7. Secondary Outcome: Oxidative Stress and Inflammatory Markers: High-sensitivity C-reactive Protein (hsCRP)
Description: high-sensitivity C-reactive protein (hsCRP)
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: 1 participant in the T1 Diabetes groups was excluded from the analysis because data was only collected in the Acipimox phase and matching Placebo data would have been required for comparison. Another participant from the Non T1D Placebo group did not have data collected.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 7
mg/L | 3.19 (3.84) | 1.98 (1.64) | 1.43 (1.11) | 1.44 (1.42)

8. Secondary Outcome: Oxidative Stress and Inflammatory Markers: Adiponectin
Description: adiponectin
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: 1 participant in the T1 Diabetes groups was excluded from the analysis because data was only collected in the Acipimox phase and matching Placebo data would have been required for comparison. Two participants (one in each of the Non-T1D study phases) did not have data collected.
Measure: Mean (Standard Deviation); unit: micrograms/mL
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 9 | 9 | 7 | 7
micrograms/mL | 11.6 (7.7) | 14.9 (10.8) | 7.3 (5.0) | 5.8 (2.1)

9. Secondary Outcome: Oxidative Stress and Inflammatory Markers: Plasminogen Activator Inhibitor (PAI-1)
Description: Plasminogen activator inhibitor (PAI-1)
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: Measure was not collected due to funding limitations.
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Heart Rate Variability
Description: Measure of autonomic function; ratio of fastest to slowest heart rate during valsalva maneuver.
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- T1D: Acipimox; No T1D: Acipimox: Drug: acipimox
  Acipimox: Subjects will take acipimox 250mg by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day.
- T1D: Placebo; No T1D: Placebo: Drug: Placebo
  Placebo: Subjects will take placebo by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day
Arm/Group | T1D: Acipimox | T1D: Placebo | No T1D: Acipimox | No T1D: Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 8
ratio | 1.37 (.17) | 1.43 (.14) | 1.59 (.19) | 1.69 (.30)

11. Secondary Outcome: Arterial Stiffness (PWV)
Description: Pulse wave velocity by Sphygmacor as a measure of aortic stiffness in m/sec. Higher values reflect a stiffer vasculature.
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: 1 participant in the T1 Diabetes groups was excluded from the analysis because data was only collected in the Acipimox phase and matching Placebo data would have been required for comparison. Additionally, one participant in each of the T1D study phases did not have data collected.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | T1D: Acipimox | T1D: Placebo | No T1D: Acipimox | No T1D: Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
m/sec | 9.24 (2.46) | 9.91 (3.30) | 6.97 (1.71) | 7.4 (1.00)

12. Secondary Outcome: Arterial Stiffness (AI)
Description: Augmentation index by Sphygmacor is a measure of aortic arterial stiffness. AI@75 is the ratio of augmented pressure/pulse pressure adjusted to a heart rate of 75.
  Higher values indicate stiffer vessels
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | T1D: Acipimox | T1D: Placebo | No T1D: Acipimox | No T1D: Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 8
ratio | 21.4 (8.4) | 19.7 (10.0) | 11.1 (13.0) | 12.4 (12.7)

13. Secondary Outcome: Metabolic Markers: Continuous Glucose Monitoring Measures
Description: Continuous glucose monitoring measures for 3 days before clamp. Collected for participants with T1 Diabetes only.
Time Frame: day 6 to 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: 1 participant was excluded from the analysis because data was only collected in the Acipimox phase and matching Placebo data would have been required for comparison.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | T1D: Acipimox | T1D: Placebo
Number analyzed (Participants) | 9 | 9
mmol/L
  Average Glucose | 8.82 (1.2) | 9.09 (0.72)
  Glycemic Variability | 3.64 (0.92) | 3.64 (0.66)

14. Secondary Outcome: Metabolic Markers: Mean 24 Hour Triglyceride and Glucose Levels
Description: mean glucose and triglycerides for the 24 hours before the 2nd overnight stay from 22 hourly measurements over 24 hours (except 0100 and 0300).
Time Frame: day 6 to 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 8
mg/dL
  glucose | 135 (28) | 131 (31) | 87 (10) | 89 (8)
  triglycerides | 59 (29) | 68 (33) | 67 (20) | 83 (27)

15. Secondary Outcome: Metabolic Markers: Insulin
Description: mean insulin for the 24 hours before the 2nd overnight stay from 22 hourly measurements over 24 hours (except 0100 and 0300).
Time Frame: day 6 to 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Measure: Mean (Standard Deviation); unit: microIU/mL
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 8
microIU/mL | 48 (25) | 47 (26) | 20 (6) | 21 (10)

16. Secondary Outcome: Metabolic Markers: Glycerol
Description: mean glycerol for the 24 hours before the 2nd overnight stay from 22 hourly measurements over 24 hours (except 0100 and 0300).
Time Frame: day 6 to 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Measure: Mean (Standard Deviation); unit: micromoles/L
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 8
micromoles/L | 86 (25) | 75 (20) | 63 (12) | 69 (14)

17. Secondary Outcome: Vascular Markers
Description: endothelin 1 measured as a marker of vascular damage
Time Frame: day 6 to 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: 1 participant in the T1 Diabetes groups was excluded from the analysis because data was only collected in the Acipimox phase and matching Placebo data would have been required for comparison. in addition, the last nonDM subjects did not have this collected due to funding limitations and futility based on prior results.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 9 | 9 | 6 | 6
pg/mL | 4.92 (1.56) | 4.9 (0.91) | 4.83 (0.92) | 4.12 (1.00)

18. Other Pre Specified Outcome: Other Mitochondrial Measures: Mito Content and Electron Transport Chain Complexes
Description: Mito content and electron transport chain complexes by western blot analysis.
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: Originally described as secondary but were actually exploratory. Not done due to funding and tissue limitations.
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Other Pre Specified Outcome: Oxidative Stress and Inflammatory Markers: Exploratory (Not Collected)
Description: thiobarbituric acid reactive substances (TBARs), glutathione disulfide (GSSG): reduced Glutathione (GSH) ratio; amplex red assay of hydrogen peroxide (H2O2) production,
Time Frame: day 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: These oxidative stress and inflammatory markers were collected, but assays were found to be unreliable. These measurements were originally erroneously described as secondary outcome measures, but are exploratory.
Arm/Group | Acipimox | Placebo
Number analyzed (Participants) | 0 | 0

20. Other Pre Specified Outcome: Counterregulatory Hormones
Description: Planned glucagon and cortisol as a markers of counteregulation, but not done due to financial limitations
Time Frame: day 6 to 7 of each of the 2 random order intervention phases; max 16 weeks post enrollment
Population: 1 participant in the T1 Diabetes groups was excluded from the analysis because data was only collected in the Acipimox phase and matching Placebo data would have been required for comparison. Incorrectly listed as secondary outcome. This was an exploratory outcome.
Arm/Group | T1 Diabetes, Acipimox | T1 Diabetes, Placebo | No T1 Diabetes, Acipimox | No T1 Diabetes, Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to about Week 16
Groups:
- T1 Placebo; No T1 Placebo: Drug: Placebo
  Placebo: Subjects will take placebo by mouth four times a day for a total of seven days plus one dose the morning of the final study visit day
Arm/Group | T1 Diabetes, Acipimox | T1 Placebo | No T1 Diabetes, Acipimox | No T1 Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/9 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T1 Diabetes, Acipimox (N=10) | T1 Placebo (N=9) | No T1 Diabetes, Acipimox (N=8) | No T1 Placebo (N=8)
bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was stopped early for two reasons: one was the serious adverse event and the other was the fact that the fatty acid lowering effect of acipimox was more short-lived than expected and we did not see the intended overall fatty acid lowering.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes